CLINICAL TRIAL: NCT07034508
Title: An Open-Label, Multicentre, Randomized Phase II Non-Inferiority Trial Comparing 4 vs 6 Cycles of CHP (21-Day Intervals) Both Combined With 6 Cycles of Polatuzumab Vedotin and Rituximab in Previously Untreated Diffuse Large B-Cell Lymphoma Patients With IPI 0-1
Brief Title: A Phase II Trial of 4 vs 6 Cycles of CHP Combined With Polatuzumab Vedotin-Rituximab in Untreated DLBCL Patients With IPI 0-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025053
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4×Pola-RCHP followed by 2×Pola-R (Experimental): Participants will receive:
  Polatuzumab Vedotin: 1.8 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1 of every cycle for 6 cycles.
  Rituximab: 375 milligrams per square meter (mg/m^2) IV on Day 1 of every cycle for 6 cycles.
  Cyclophosphamide: 750 mg/m^2 IV on Day 1 of every cycle for 4 cycles. Doxorubicin: 50 mg/m^2 IV on Day 1 of every cycle for 4 cycles. Prednisone: 100 milligrams per day (mg/day) orally (PO) on Days 1-5 of each 21-day cycle for 4 cycles.
  This Pola-RCHP regimen is repeated for 4 cycles, followed by 2 cycles of Polatuzumab Vedotin and Rituximab.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone
- 6×Pola-RCHP (Active Comparator): Participants will receive:
  Polatuzumab Vedotin: 1.8 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1 of every cycle for 6 cycles.
  Rituximab: 375 milligrams per square meter (mg/m^2) IV on Day 1 of every cycle for 6 cycles.
  Cyclophosphamide: 750 mg/m^2 IV on Day 1 of every cycle for 6 cycles. Doxorubicin: 50 mg/m^2 IV on Day 1 of every cycle for 6 cycles. Prednisone: 100 milligrams per day (mg/day) orally (PO) on Days 1-5 of each 21-day cycle for 6 cycles.
  This regimen is repeated for 6 cycles
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Rituximab — Rituximab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.

SUMMARY:
This is an open-label, multicentre, randomized phase II non-inferiority trial aiming to compare the efficacy and safety of 4 versus 6 cycles of CHP (administered at 21-day intervals), both in combination with 6 cycles of polatuzumab vedotin and rituximab, in previously untreated patients with diffuse large B-cell lymphoma (DLBCL) and an International Prognostic Index (IPI) score of 0-1. The study's primary objective is to determine if shorter CHP duration can achieve comparable outcomes to the standard 6-cycle regimen when combined with polatuzumab vedotin and rituximab

DETAILED DESCRIPTION:
The POLARIX study demonstrated that the Pola-R-CHP regimen (replacing vincristine in R-CHOP with Pola) significantly improves progression-free survival (PFS) and is safer than traditional R-CHOP. The FLYER study suggested that 4 cycles of R-CHOP followed by 2 additional doses of rituximab in young, low-risk DLBCL patients (IPI 0-1) are as effective as 6 cycles of R-CHOP and result in lower toxicity. Based on the efficacy of Pola-R-CHP and the potential for reducing treatment intensity in low-risk patients, this study will evaluate whether 4 cycles of Pola-R-CHP followed by 2 cycles of Pola-R are non-inferior to 6 cycles of Pola-R-CHP in treatment-naive low-risk DLBCL patients (IPI 0-1), with a potentially better safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, untreated, biopsy-proven CD20 positive diffuse large B-cell lymphoma (DLBCL)
* Age ≥18yo and ≤80yo at the time of signing consent
* International Prognostic Index (IPI) score 0-1
* ECOG 0-2
* Have measurable disease on a pre-chemotherapy PET/CT, defined as at least one bi-dimensionally measurable nodal lesion of >1.5cm in longest dimension, or at least one bi-dimensionally measurable extranodal lesion of >1.0cm in longest dimension
* Life expectancy greater than or equal to (>/=)12 months
* Left ventricular ejection fraction (LVEF) >/= 50 percent (%) on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematologic function
* Female participants: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods and refrain from donating eggs.
* Male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom and agreement to refrain from donating sperm.

Exclusion Criteria:

* Patients with central nervous system or primary mediastinal lymphoma, and patients with transformed lymphoma.
* Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, severe infectious diseases, etc.
* Pregnant or lactating women.
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV; positive by RNA polymerase chain reaction [PCR]) infection.
* Patients with concurrent other tumors or a history of tumors, or who have received anti-tumor treatment (including major surgery) within the last 4 weeks.
* Allergic reactions to polatuzumab vedotin.
* Other conditions where the investigator deems the patient ineligible for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) | up to the end of 6 cycles of treatment (each cycle is 28 days)]
  To assess the complete response rate (CR) at the end of treatment with Treatment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to the end of 6 cycles of treatment (each cycle is 28 days)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment
Duration of Response (DoR) | up to 2 years
  The length of time between the achievement of criteria for response to treatment (first documented complete or partial response) and the first documented relapse or progression.
Progression-free survival (PFS) | up to 2 years
  The time from the enrollment of a subject to the occurrence of (in any way) progression of disease or Death for any reason. patients with indeterminate recurrence or Death at the last follow-up, defined as the date of the last Investigation
To identify biomarkers | up to 2 years
  To identify biomarkers that may predict response to a combination regimen, biomarkers associated with progression to a more severe disease state, biomarkers that are sensitive to the development of Adverse event, biomarkers that provide evidence of the activity of the combination, or biomarkers that may enhance the understanding or understanding of the biology of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- China Institute of Hematology and Blood Diseases Hospital, Tianjin, China